CLINICAL TRIAL: NCT04054167
Title: Phase II Trial to Assess the Efficacy of Ultra Low Radiation Dose Delivered Prior or After Chemotherapy Free Targeted Therapy for the Treatment of Relapsed/Refractory Mantle Cell Lymphoma
Brief Title: Ultra Low Dose Radiation Delivered Before or After Chemotherapy-Free Targeted Therapy in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0348; NCI-2019-01729 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0348 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-07-02; First posted 2019-08-13 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ultra low dose radiation therapy) (Experimental): Patients undergo ultra low dose radiation for 1-2 days before chemotherapy free-targeted therapy. Patients may receive a second, longer course of radiation if the lesion treated does not respond.
  Interventions: Drug: Low Dose Radiation Therapy

INTERVENTIONS:
Drug: Low Dose Radiation Therapy — Undergo ultra low dose radiation
  Other Names: Low Dose Radiation

SUMMARY:
This phase II trial studies how well ultra low dose radiation works before or after chemotherapy-free targeted therapy in treating patients with mantle cell lymphoma that has come back or does not respond to treatment. Radiation therapy uses high energy x-rays to kill cancer cells and shrink tumors. Ultra low dose radiation is generally associated with a lower risk of side effects which may allow patients to be able to receive low-dose radiation therapy more often than high-dose radiation therapy. This trial may help doctors learn if giving ultra low dose radiation helps control mantle cell lymphoma and improves response to chemotherapy free targeted therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of adding ultra low dose radiation (ULDR) to chemotherapy free-targeted therapy (CTFTT) in contributing to a durable overall response in treated locations by estimating overall response rate (ORR) at 3 months.

SECONDARY OBJECTIVES:

I. To evaluate if ULDR can improve progression-free survival and overall survival.

II. To evaluate the prognostic factors associated with inferior progression-free survival, including patient related and previous treatment related and if radiation can overcome these prognostic factors.

III. To evaluate if radiation helps to bridge patients to other investigational drugs, by decreasing the disease bulk, controlling their symptoms, and maintaining a good performance status.

OUTLINE:

Patients undergo ultra low dose radiation for 1-2 days before chemotherapy free-targeted therapy. Patients may receive a second, longer course of radiation if the lesion treated does not respond.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed diagnosis of mantle cell lymphoma with positivity in tissue biopsy. Biopsy does not need to be done of the lesions to be treated.
* Patients can be newly diagnosed or previously treated relapsed and/or refractory MCL.
* Understand and voluntarily sign an IRB-approved informed consent form.
* Age ≥ 18 years at the time of signing the informed consent.
* Patients must have bi-dimensional measurable disease (Measurable disease by CT scan defined as at least 1 lesion that measures =/>1.5 cm in single dimension.) Patient presenting with lesions in the presence of leukemia phase (peripheral blood involvement), non-measurable disease, gastrointestinal (GI) MCL, or bone marrow (BM) MCL are also eligible.
* Gastrointestinal or bone marrow or spleen only patients are allowable and will be analyzed separately.
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less (see Appendix 1).
* Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty.
* Females of childbearing potential (FCBP)1 must have a negative serum or urine pregnancy test and must be willing to use acceptable methods of birth control during the study and for 30 days after the last dose of study treatment.
* Male patients must use an effective barrier method of contraception during the study and for 30 days following the last dose of study treatment if sexually active with a female of childbearing potential.
* Serum bilirubin <1.5 mg/dl and Cr Clearance ≥ 30 mL/min, platelet count >25,000/mm3 and absolute neutrophil count (ANC) > 1,000/mm3, AST (SGOT) and ALT (SGPT) < 3 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present.
* Patients who have bone marrow infiltration by MCL are eligible if their ANC is ≥ 1000/mm3 [growth factor not allowed] or their platelet level is ≥ 25,000/mm3

Exclusion Criteria:

* Has had prior radiation therapy to the potential radiation target such that additional radiation therapy is considered unsafe by the treating radiation oncologist
* Has a diagnosis of active scleroderma or lupus or any other autoimmune disease that by the opinion of the treating radiation oncologist would put the patient at unacceptable risk of toxicity.
* Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled infection, active/symptomatic coronary artery disease, COPD, renal failure, active hemorrhage, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk and would prevent the subject from signing the informed consent form.
* Pregnant or breast-feeding females.
* All patients with central nervous system lymphoma that needs attention prior to treatment of the lesions.
* If the total fields of radiation will include a marrow volume of more than 40%. Physician can include as many fields to respect the 40 % of marrow volume and come back in 4-6 weeks later to address the rest of the disease after insuring that the Blood counts are adequate. Blood counts should be back to back to the numbers prior to starting the first phase of radiation +- 10% variance.
* If given radiation prevent them from going through an alternative phase I trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | At 3 months
  ORR will be based on the tumors residing within the radiated field using the sum of the longest tumoral axes treated. Responses are defined as follows: i) complete response (CR): > 75% reduction in the sum of the longest tumoral axes treated within a radiation field; ii) partial response (PR): 50 to 75% reduction; and stable disease (SD): a reduction < 50%. Progressive disease will be defined as any relative increase in the sum of the longest tumoral axes within the radiated field. ORR will be assessed by positron emission tomography (PET)/computed tomography (CT) at 3-months after the conclusion of ultra low dose radiation (ULDR). The Lugano Classification will be used to assess tumor response. Will estimate ORR at 3 months by providing an exact 95% confidence interval for the evaluable study population.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the start of ULDR treatment to the time of a progression or death, assessed up to 5 years
  Will be estimated at select time points of interest using the Kaplan-Meier method for all patients enrolled in the study. The origination point for time will begin at the inception of ULDR. Cox proportional hazards regression will be used to evaluate potential prognostic factors.
Overall survival | From the start of ULDR treatment to the time of death or loss to follow-up, assessed up to 5 years
  Will be estimated at select time points of interest using the Kaplan-Meier method for all patients enrolled in the study. The origination point for time will begin at the inception of ULDR. Cox proportional hazards regression will be used to evaluate potential prognostic factors.
ATM mutational status | At 3 months
  Logistic regression will be utilized to assess the effect of patient characteristics such as ATM mutational status, on the Overall Response Rate(ORR ).
PET/CT metabolic parameters | At 3 months
  Logistic regression will be utilized to assess the effect of patient characteristics such PET/CT metabolic parameters, on the Overall Response Rate (ORR).
The Descriptive Statistics of Patient Characteristics of the Transitions to other Investigational Drugs. | Up to 5 years
  Will be used to summarize patient characteristics such as transitions to other investigational drugs at select time points in a patient's follow-up domain. These summaries will indicate if ULDR helps to bridge patients to other investigational drugs, by decreasing the disease bulk, controlling their symptoms, and maintaining a good performance status.
The Descriptive Statistics of Patient Characteristics of the Patients Disease Bulk. | Up to 5 years
  Will be used to summarize patient characteristics such as disease bulk at select time points in a patient's follow-up domain. These summaries will indicate if ULDR helps to bridge patients to other investigational drugs, by decreasing the disease bulk, controlling their symptoms, and maintaining a good performance status.
The Descriptive Statistics of Patient Characteristics of the Patients Symptoms. | Up to 5 years
  Will be used to summarize patient characteristics such as symptoms at select time points in a patient's follow-up domain. These summaries will indicate if ULDR helps to bridge patients to other investigational drugs, by decreasing the disease bulk, controlling their symptoms, and maintaining a good performance status.
The Descriptive Statistics of Patient Characteristics of the Patients Performance status | Up to 5 years
  Will be used to summarize patient characteristics such as performance status at select time points in a patient's follow-up domain. These summaries will indicate if ULDR helps to bridge patients to other investigational drugs, by decreasing the disease bulk, controlling their symptoms, and maintaining a good performance status.

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org